CLINICAL TRIAL: NCT01191034
Title: Phase I/II Study of Peptide Vaccination Associated With Tumoral Immunomodulation With Proinflammatory Cytokines and Imiquimod in Patients With Advanced Metastatic Melanoma
Brief Title: Peptide Vaccination Associated With Tumoral Immunomodulation in Patients With Advanced Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Completion after 2 patients then stop due to end of validity of vaccine peptide
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Luc 10-002
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vaccine MAGE-3.A1 peptide, or the NA17.A2 peptide + IL-2, IFN-α and GMCSF, Imiquimod. — The vaccine will be either the MAGE-3.A1 peptide, or the NA17.A2 peptide, or both,matching the patient's HLA type and the gene expression of his tumor. If both antigens are expressed, then the patient will receive both peptides.
  This treatment will combine subcutaneous peritumoral injections of IL-2, IFN-α and GMCSF,as well as topical applications of imiquimod.

SUMMARY:
Human cancers express tumor antigens that can be targeted by cytolytic T lymphocytes (CTL). These antigens consist of a small peptide, derived from endogenous proteins, that is presented at the cancer cell's surface by an HLA class I molecule. Such antigenic peptides, including MAGE-3.A1 and NA17.A2, have been tested in experimental therapeutic vaccines to elicit CTL responses in cancer patients, mainly with metastatic melanoma. Up to now, only rare tumor responses have been observed.

Tumor resistance to CTL killing is the most likely explanation for the poor effectiveness of cancer vaccines. This resistance is probably acquired by the tumor during its development and selected by its repetitive challenge with spontaneous anti-tumoral immune responses. The precise molecular mechanisms of tumor resistance remain unknown. The observation that tumor-infiltrating lymphocytes (TIL) purified from melanoma metastases can recognize and kill autologous tumor cells in vitro, whilst they seem unable to control tumor growth in vivo, suggests that this resistance is hosted by the tumor environment, rather than being the result of a generalized immune suppression.

The investigators have developed a murine model of cutaneous graft rejection that mimics the situation in melanoma. Female CBA mice do not reject syngeneic male skin grafts, even though they mount a spontaneous CTL response against H-Y, a male specific minor histocompatibility antigen, following grafting. The investigators have tested various experimental procedures aimed at inducing effective graft rejection in these mice. This was obtained with a combination of IFN-α, IL-2, GM-CSF, each administered separately under the skin graft, associated with topical applications of imiquimod. All these agents are available as registered drugs. Based on this murine model of cutaneous allograft rejection, the investigators postulate that local immunomodulation with this combination can trigger an effective tumor rejection process, and induce a more efficient and long-lasting anti-tumoral immune response following peptide vaccination.

DETAILED DESCRIPTION:
Patients will receive the following treatments:

1. Vaccinations:

   The vaccine will be the MAGE-3.A1 and/or the NA17.A2 peptide, matching the patient's HLA type and the gene expression of his tumor. If both antigens are expressed, then the patient will receive both peptides.
2. Local treatment with a combination of immunomodulatory drugs:

This treatment will combine peritumoral injection of IL-2, IFN-α and GM-CSF (6000 IU, 100.000 IU and 300 ng per tumor injected, respectively), as well as topical application of imiquimod (applied during 24h). The peritumoral injections of cytokines will be given on days +2,+3,+4,+7,+8 and +9, and the Aldara® cream will be applied on days +2 and +7 following vaccines 3 and 4. One or 2 cutaneous lesions will be treated, if there are 2 or more such lesions present at day 29 of the treatment, respectively.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with histologically proven cutaneous melanoma at one of the following AJCC stages.Regional metastatic disease (any T; N2c or N3; M0). Distant metastatic disease (any T; any N; M1a, M1b or M1c*).*except uncontrolled brain metastasis.
* 2. HLA-A1 or HLA-A2 (by serology or molecular biology).
* 3. MAGE-3 gene expression by the tumor if patient is HLA-A1 and/or NA17 gene expression by the tumor if patient is HLA-A2 (determined by RT-PCR analysis).
* 4. Measurable Disease (RECIST v1.1)Patients must have at least 2 cutaneous metastases, suitable for peri-tumoral injection and surgical resection, with their largest diameter equal to or greater than 5 mm.
* 5. Age ≥ 18 years.
* 6. Karnosky Performance status (KPS) ≥70 or WHO performance status of 0 or 1
* 7. Expected survival of at least 6 months.
* 8. Normal laboratory values : Platelet count ≥100x103/μL,Leucocyte count ≥ 3x103/μL, Hemoglobin ≥ 9 g/dL, ASAT and ALAT ≤ 2xUNL, Serum creatinine ≤1.5xUNL, Total bilirubin ≤ 1.5xUNL, LDH ≤ 1.5xUNL
* 9. Viral serology : negative antibodies for HCV & HIV; negative antigens for HBV.
* 10. Patient should agree to perform biopsies and blood collections for translational research.
* 11. Signed informed consent from the patient or legal representative must be obtained.

Exclusion Criteria:

1. Uncontrolled brain or central nervous system metastases.
2. Previous treatment for the melanoma within 6 weeks from inclusion, with any reagent known to modulate the immune system such as a cancer vaccine, interferon-alpha, interleukins or anti-CTLA-4 antibodies.
3. Previous chemotherapy, radiotherapy, corticotherapy, or other immune suppressive therapy within 4 weeks from inclusion.
4. Clinically significant cardiovascular disease (including cardiac insufficiency NYHA grade III and IV, unstable angina, arrythmia, myocardial infarction, symptomatic congestive heart failure) in the past 12 months before enrollment.
5. Other serious acute or chronic illnesses, e.g. active infections requiring antibiotics, bleeding disorders or other conditions requiring concurrent medications not allowed during this study.
6. Other malignancy within 3 years prior to entry in the study, except for treated non-melanoma skin cancer and in situ cervical carcinoma.
7. Active immunodeficiency disease or autoimmune disease (Vitiligo is not an exclusion criterion).
8. Lack of availability for immunological and clinical follow-up assessments.
9. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
10. Subject pregnant or breastfeeding, or planning to become pregnant within 6 months after the end of treatment.
11. Subject (male or female) not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months after the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08-01 (Actual)

PRIMARY OUTCOMES:
To determine whether peptide vaccination associated with local peritumoral treatment with a combination of interleukin-2, interferon-alpha, granulocyte-macrophage colony stimulating factor, and imiquimod, induces tumor responses. | week 11 day 71
  Tumor response will be assessed in accordance with the Modified RECIST version 1.1

SECONDARY OUTCOMES:
To document the toxicity of treatment | at each visit
  Laboratory tests, vital sign measurements, physical exams and patient queries will be performed to detect new abnormalities and deteriorations of any pre-existing conditions.
  All clinically significant abnormalities and deteriorations should be recorded in the Case Report Forms as Adverse Events and graded according to the National Cancer Institute CTCAE v3.0.
To document whether this association induces cytolytic T lymphocyte responses to the vaccine antigens | at week 11, day 71
  CTL responses will be assessed by comparing either the anti-MAGE-3.A1 or the anti- NA17.A2 CTLp frequency in the pre- and post-immune blood of patients vaccinated with the respective antigen.

CONTACTS AND LOCATIONS:
Overall Officials: Baurain Jean-Francois, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No